CLINICAL TRIAL: NCT04195191
Title: Effectiveness of an Intervention to Improve the Adherence to Treatment of New Medicines From the Community Pharmacy
Brief Title: Intervention to Improve the Adherence in Community Pharmacies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Andalusian School of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2018713122010
Record Dates: First submitted 2018-10-17; First posted 2019-12-11 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2019-12

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD; Arterial Hypertension; Diabetes Mellitus
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypertension; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: cluster randomized controlled trial.
Who Masked: Outcomes Assessor
Masking Description: The statistical analysis will be performed by a person who would be blinded to which arm were assigned the subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): The usual practice by community pharmacies
  Interventions: Other: Placebo
- ANM (Experimental): This is an intervention based on pharmaceutical-patient communication through an open and fluid conversation, aimed at evaluating the patient's relationship with their new prescription, detecting possible problems, concerns and false beliefs or visual expectations.
  Interventions: Other: ANM

INTERVENTIONS:
Other: ANM — communication intervention
  Arms: ANM
Other: Placebo — regular assistance in community pharmacies
  Arms: Placebo

SUMMARY:
The ANM is the first initiative that puts advanced pharmaceutical care into practice in Andalusia (Spain). The aim of this is study is to evaluate the effectiveness of the intervention Assistance to New Medicines (ANM) in the improvement of adherence to treatment in community pharmacies.

DETAILED DESCRIPTION:
Design: parallel cluster pragmatic randomized controlled trial. The study includes patients users of a community pharmacies, who meet the following inclusion criteria: patient who starts treatment of any of the following pathologies: Chronic Obstructive Pulmonary Disease (COPD), Arterial Hypertension or Diabetes Mellitus in Andalusia (Spain).

In order to avoid possible contamination between patients assigned to the control and intervention group, randomization will be carried out at the pharmacy level; preventing the pharmacist from applying part of the intervention to the control group.

Interventions: patients randomized: (i) current practice; or (ii) ANM intervention thru a pharmacist delivered support for a newly prescribed medicine.

ELIGIBILITY:
Inclusion Criteria: patient who starts treatment of any of the following diseases:

* Chronic Obstructive Pulmonary Disease (COPD).
* Arterial Hypertension
* Diabetes Mellitus.
* Anticoagulants

Exclusion Criteria:

* those users who do not know how to read and write in Spanish,
* Suffer from a physical or mental disorder that makes it impossible to perform the

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-01-18 (Actual); Primary Completion 2020-03-02 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Adherence to treatment | Ten weeks
  adherence to treatment may be defined as the extent to which the patient's history of therapeutic drug-taking coincides with the prescribed treatment.
Adherence to treatment | Six months
  adherence to treatment may be defined as the extent to which the patient's history of therapeutic drug-taking coincides with the prescribed treatment.

SECONDARY OUTCOMES:
Satisfaction with the service | Ten weeks and six months
  The degree to which the individual regards the health care service or product or the manner in which it is delivered by the provider as useful, effective, or beneficial. The satisfaction with the service, will be collected thru a likert question (1 not satisfied, 10 very satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Andalusian School of Public Health & CIBER en Epidemiología y Salud Pública (CIBERESP)., Granada, Spain

IPD SHARING:
Plan to Share IPD: No